CLINICAL TRIAL: NCT06302400
Title: Individualized Dosimetry for Holmium-166 Radioembolization in Patients With Unresectable Hepatocellular Carcinoma; a Multi-centre, Interventional, Non-randomized, Non-comparative, Open Label, Early Phase II Study
Brief Title: Individualized Dosimetry for Holmium-166 Radioembolization in Patients With Unresectable Hepatocellular Carcinoma
Acronym: RHEPaiR
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Terumo Europe NV permanently discontinued production of Holmium platform SIRT product range
Sponsor: Imperial College London (Other)
Collaborators: Terumo Europe N.V. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RS-IC04
Record Dates: First submitted 2024-02-06; First posted 2024-03-08 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Carcinoma, Hepatocellular
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Radioembolisation with 166Holmium microspheres (Experimental)
  Interventions: Device: 166Holmium microspheres (QuiremSpheres®)

INTERVENTIONS:
Device: 166Holmium microspheres (QuiremSpheres®) — QuiremSpheres® are a biocompatible microsphere that contain the radionuclide holmium-166 (166Ho), which emits gamma-radiation (81 keV) and high-energy (1.81 MeV) beta-particles.

SUMMARY:
The goal of this clinical trial is to test the safety and effectiveness of a medical device called 166-Holmium microspheres (QuiremSpheres®) in patients with hepatocellular carcinoma (HCC) . The main questions it aims to answer are:

* What is the safety and toxicity profile of the 166-Holmium microspheres?
* Is the device effective in treating HCC?

Participants will undergo a range of screening procedures to confirm they are eligible and to record their baseline results, including:

* A Computed Tomography (CT) scan
* A Magnetic Resonance Imaging (MRI) scan
* Blood tests
* Quality of life questionnaires

Before receiving treatment with QuiremSpheres® the participant will receive a 'scout' dose of the microspheres, to check whether there is distribution of the radioactivity to other non-target areas of the body. This is measured using Single-Photon Emission Computed Tomography-CT imaging. If the distribution to non-target areas is deemed to not be too high, the participant will go on to receive the individualised therapeutic dose of QuiremSpheres®. Follow-up visits will occur 3 and 6 weeks post-treatment dose, and then at 3 and 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Provided written informed consent.
2. Female or male aged 18 years and over.
3. Diagnosis of HCC established according to AASLD criteria: nodule >1 cm in a patient at risk for HCC, with combination of arterial hypervascularity and venous or delayed phase wash-out on multiphase CT-scan or MRI-scan. LR-5 and LR- 4 based on Liver Imaging Reporting and Data System can be included.
4. No curative treatment options (resection, transplant, or in case of solitary tumour, RFA).
5. Life expectancy of at least 6 months.
6. ECOG Performance status 0-1.
7. Liver-dominant disease (maximum 5 lung nodules all ≤1.0 cm, solitary clinically stable adrenal metastasis, and mesenteric or portal lymph nodes all ≤2.0 cm are accepted).
8. Child-Pugh class A5-6 or B7.
9. At least one measurable liver lesion according to the modified RECIST criteria.
10. Negative pregnancy test for women of childbearing potential. Female patients of childbearing potential should use a highly effective acceptable method of contraception (oral contraceptives, barrier methods, approved contraceptive implant, long-term injectable contraception, intrauterine device or tubal ligation) or should be more than 1 year postmenopausal or surgically sterile during their participation in this study (from the time they sign the consent form), to prevent pregnancy.

Exclusion Criteria:

1. Evidence of significant extrahepatic disease (MRI-scan liver and multiphase abdominal CT as well as a thoracic CT are routinely performed at screening).
2. Hepatic radiation therapy within the last 4 weeks before the start of study therapy.
3. Previous or current treatment with RE. Previous treatment with TACE, surgery, RFA, and previous or current treatment with systemic treatment are allowed.
4. Major surgery within 4 weeks or incompletely healed surgical incision before starting study therapy.
5. Serum bilirubin > 34 umol/L in the absence of a reversible cause
6. Glomerular filtration rate <35 ml/min.
7. Non-correctable INR >1.5 in case of femoral approach (as opposed to radial).
8. Platelet count <50 109/l.
9. Significant cardiac event (e.g., myocardial infarction, superior vena cava (SVC) syndrome, New York Heart Association (NYHA) classification of heart disease ≥2) within 3 months before entry, or presence of cardiac disease that in the opinion of the investigator increases the risk of ventricular arrhythmia.
10. Pregnancy or breastfeeding.
11. Patients suffering from psychic disorders that make a comprehensive judgment impossible, such as psychosis, hallucinations and/or depression.
12. Patients who are declared incapacitated.
13. Previous enrolment in the present study.
14. Male patients who are not surgically sterile or do not use an acceptable method of contraception during their participation in this study (from the time they sign the consent form), to prevent pregnancy in a partner.
15. Evidence of untreated, clinically significant grade 3 portal hypertension (i.e. large varices at oesophagi-gastro-duodenoscopy). In these cases, therapy with non-selective beta-blocker (propranolol) or rubber band ligation should be instituted according to accepted guidelines. In case of small varices, prophylactic propranolol is advised.
16. Portal vein thrombosis (tumour and/or bland) of the main branch (diagnosed on contrast enhanced transaxial images). Involvement of the right or left portal vein branches and more distal is accepted.
17. Untreated active hepatitis. In case of detectable viral HBV load, appropriate treatment should be instituted.
18. Transjugular intrahepatic portosystemic shunt (TIPS).
19. Body weight over 150 kg (because of maximum table load).
20. Severe allergy for intravenous contrast used (Visipaque®)
21. Lung shunt >30 Gy, as calculated using scout dose SPECT/CT.
22. Extrahepatic deposition of scout dose activity. Activity in the falciform ligament, portal lymph nodes and gallbladder is accepted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2024-02-22 (Actual); Primary Completion 2025-03-04 (Actual); Study Completion 2025-03-04 (Actual)

PRIMARY OUTCOMES:
The incidence of adverse and serious adverse events in patients receiving individualized treatment with 166Ho- microspheres, using National Cancer Institute CTCAE v5.0. | Approximately 8 months

SECONDARY OUTCOMES:
The rate of efficacy as defined as overall response rate (ORR) in patients receiving individualized treatment with 166Ho- microspheres, using modified RECIST (mRECIST) response evaluation criteria. | Approximately 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Rohini Sharma, Professor, Principal Investigator — Imperial College London
Locations (1):
- Imperial College Healthcare NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Qurashi M, Martinez M, Ward C, Wyard C, Izadi H, Bowen C, Khan SR, Tait P, Smits M, de Bruijne J, Thomas R, Lam MGEH, Sharma R. Individualised dosimetry for holmium-166 RE in patients with unresectable hepatocellular carcinoma; a multi-centre, interventional, non-randomised, non-comparative, open label, phase II study: RHEPaiR. BMJ Open. 2025 Nov 19;15(11):e097066. doi: 10.1136/bmjopen-2024-097066. PMID 41263849